CLINICAL TRIAL: NCT00894335
Title: Anesthesiological Management of Hemodynamics and Gas Exchange for Retroperitoneal Adrenalectomies
Brief Title: Anesthesia Management of Retroperitoneal Adrenalectomies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Harald Groeben, Prof. Dr., Department of Anesthesiology and CCM , Clinics Essen-Mitte
Other Study IDs: retroper adrenal
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2009-05

CONDITIONS: Adrenal Tumors
Keywords: retroperitoneoscopic adrenalectomy; intraoperative arterial-alveolar Carbon dioxide Difference
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Pheochromocytoma
- 2: Conn-Syndrome
- 3: Cushing disease
- 4: Metastasis
- 5: Non-functional tumor

SUMMARY:
This study is a prospective, perioperative evaluation of hemodynamic and respiratory parameters in patients undergoing retroperitoneoscopic adrenalectomies.

DETAILED DESCRIPTION:
Due to their underlying disease, patients with adrenal tumors are prone to episodes of hyper- and hypotension. Furthermore, excessive hypercarbia and an increased arterial-alveolar CO2 difference can be seen during these operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an adrenal tumor

Exclusion Criteria:

* Age below 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adrenal tumors scheduled for retroperitoneal adrenalectomies
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-05; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Arterial-alveolar Carbon dioxide Difference | 3 years

SECONDARY OUTCOMES:
Perioperative maximal mean arterial pressure | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Harald Groeben, Prof, M.D., Principal Investigator — Clinics Essen-Mitte
Locations (1):
- Clinics Essen-Mitte, Essen, Germany

REFERENCES:
- [Background] Walz MK, Alesina PF, Wenger FA, Deligiannis A, Szuczik E, Petersenn S, Ommer A, Groeben H, Peitgen K, Janssen OE, Philipp T, Neumann HP, Schmid KW, Mann K. Posterior retroperitoneoscopic adrenalectomy--results of 560 procedures in 520 patients. Surgery. 2006 Dec;140(6):943-8; discussion 948-50. doi: 10.1016/j.surg.2006.07.039. PMID 17188142